CLINICAL TRIAL: NCT02933853
Title: This Trial is Conducted in Europe. The Aim of This Trial is to Investigate Pharmacokinetic (the Exposure of the Trial Drug in the Body) and Pharmacodynamic (the Effect of the Investigated Drug on the Body) Properties of Faster-acting Insulin Aspart in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Trial Investigating the Pharmacokinetic and Pharmacodynamic Properties of Faster-acting Insulin Aspart in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-4265; 2016-000200-28 (EudraCT Number); U1111-1178-3964 (Other: WHO)
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Faster Aspart (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- Insulin Aspart (Active Comparator)
  Interventions: Drug: Insulin Aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — A single dose administered subcutaneously (s.c., under the skin). The dose level will be 0.3 U/kg body weight.
  Arms: Faster Aspart
Drug: Insulin Aspart — A single dose administered subcutaneously (s.c., under the skin). The dose level will be 0.3 U/kg body weight.
  Arms: Insulin Aspart

SUMMARY:
A Trial Investigating the Pharmacokinetic and Pharmacodynamic Properties of Faster-acting Insulin Aspart in Subjects with Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent. The total number of subjects aged 65-75 years (both inclusive) must NOT exceed 25.
* Subjects diagnosed (clinically) with type 2 diabetes mellitus for at least 12 months (365 days) prior to the day of screening
* HbA1C below or equal to 9.5 % based on central laboratory analysis

Exclusion Criteria:

* Smoker (defined as a subject who is smoking more than one cigarette or the equivalent per day) who is not able or willing to refrain from smoking and use of nicotine substitute products during the in-patient period
* Surgery or trauma with significant blood loss (more than 500 mL) within the last 90 days prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0 to 30 minutes

SECONDARY OUTCOMES:
Maximum observed serum insulin aspart concentration | Within 0 to 12 hours after dosing
Area under the glucose infusion rate curve | From 0 to t, where t is the last time where glucose infusion rate (GIR) exceeds zero (within 0 to 12 hours after dosing)
Maximum glucose infusion rate | Within 0 to 12 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Result] Pieber TR, Svehlikova E, Brunner M, Halberg IB, Due Thomsen KM, Haahr H. Fast-acting insulin aspart in people with type 2 diabetes: Earlier onset and greater initial exposure and glucose-lowering effect compared with insulin aspart. Diabetes Obes Metab. 2019 Sep;21(9):2068-2075. doi: 10.1111/dom.13767. Epub 2019 Jun 10. PMID 31069935